CLINICAL TRIAL: NCT04464408
Title: A Trial of Favipiravir Therapy in Adults With Mild Coronavirus Disease COVID-19
Brief Title: Favipiravir Therapy in Adults With Mild COVID-19
Acronym: Avi-Mild
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC 20/220/R
Record Dates: First submitted 2020-06-28; First posted 2020-07-09 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Favipiravir; COVID19; Mild illness; Saudi Arabia
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental): Favipiravir: 1800 mg (9 tablets) by mouth twice daily for one day, followed by 800mg (4 tablets) twice daily (Maximum days of therapy is 7 days)
  Interventions: Drug: Favipiravir
- Placebo (Placebo Comparator): 9 tablets by mouth twice daily for one day, followed by 4 tablets twice daily (Maximum days of therapy is 7 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Favipiravir — 1800 mg twice daily for one day, followed by 800mg (4 tablets) twice daily
  Arms: Favipiravir
Drug: Placebo — (9 tablets) by mouth twice daily for one day, followed by (4 tablets) twice daily (Maximum days of therapy is 7 days)
  Arms: Placebo

SUMMARY:
Favipiravir is a selective and potent inhibitor of inﬂuenza viral RNA polymerase. It acts as a purine analogue, which selectively inhibits viral RNA-dependent RNA polymerase (RdRps). It has the characteristic of acting on RNA viruses including Ebola and Coronaviruses especially novel coronavirus (2019-nCoV). The purpose of this study is to evaluate the clinical efficacy and safety of Favipiravir in comparison to placebo in the treatment of mild COVID-19 cases. It is a Multicenter, randomized double-blinded, parallel-group trial.

ELIGIBILITY:
Inclusion Criteria

Patients must be eligible according to the following criteria for enrollment

1. Should be at least 18 years of age
2. Male or non-pregnant female (pregnancy testing is not mandatory. If the patient requests or is not sure, the study team will provide it)
3. Diagnosed with mild COVID-19* confirmed by positive PCR test for SARS-CoV-2 at the time of recruitment, a result within the last five days
4. Patients have to be enrolled within 5 days of disease onset.

Exclusion criteria

Patients meeting any of the following criteria will be excluded from trial enrolment:

1. Patients with concomitant documented bacterial pneumonia established through positive sputum cultures
2. Patients who are pregnant or breastfeeding
3. Known sensitivity/allergy to Favipiravir (If Faviparavir was used for COVID-19 in the patient previously for influenza)
4. Major comorbidities increasing the risk of study drug including

   * Hematologic malignancy
   * Advanced (stage 4-5) chronic kidney disease or dialysis therapy
   * Severe liver damage (Child-Pugh score C, AST> 5 times the upper limit)
   * HIV
   * Gout/history of Gout or hyperuricemia (two times above the ULN)

(6) Having used Favipiravir or participated in any other interventional drug clinical study within 30 days before the first dose of study drug (i.e., the patient received it for influenza previously) (7) The investigator believes that participating in the trial is not in the best interests of the patient, or the investigator considers unsuitable for enrollment (such as unpredictable risks or subject compliance issues) (8) Clinical prognostic non-survival, palliative care, or in a deep coma and have no response to supportive treatment within three hours of admission.

(9) Hospitalized patients for mild, moderate, or severe COVID-19

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
PCR negative | 15 days
  Time from randomization to negativity in RT-PCR nucleic acid test for COVID-19 within 15 days of randomization

SECONDARY OUTCOMES:
Time from randomization to clinical recovery | 15 days
  The duration from start of treatment (Favipiravir or placebo) to normalization of pyrexia, respiratory symptoms, and relief of cough (or other relevant symptoms at enrollment) that is maintained for at least 72 hours.
Evaluate symptoms progression | 28 days
  Evaluate symptoms severity and the disease course progression in both arms till 28 days after starting the medicine.
Evaluate Faviparivirs effect | 15 days
  To evaluate Favipiravir's effect on the requirement of the use of antipyretics, analgesics, or antibiotics within 15 days after starting medicine.
Evaluate Favipiravir's effect | 28 days
  To evaluate Favipiravir's effect on disease complications within 28 days after starting medicine (hospitalization, ICU admission, or Mechanical ventilation )
Evaluate the safety of Favipiravir | 28 days
  Evaluate the safety of investigational drug compared to the control arm within 15 days after starting the medicine. This is assessed by allergic reactions, medication intolerance, liver toxicity, and hyperuricemia in subjects

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bosaeed, Principal Investigator — KAMC-RD, Ministry of National Guard Health Affairs (MNGHA), Saudi Arabia
Locations (7):
- Saudi Arabia (7):
  - King Fahad Hospital - Madinah, Al Madīnah
  - Primary Health Care-Safiyah, Al Madīnah
  - Prince Mohammed Bin Abdul Aziz Hospital - Al Madinah, Al Madīnah
  - King Abdullah Medical City - Makkah, Mecca
  - King Abdulaziz Medical City - Riyadh, Riyadh
  - Primary Health Care-Al Mansoura, Riyadh
  - Primary Health Care-Al Urijah, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosaeed M, Alharbi A, Hussein M, Abalkhail M, Sultana K, Musattat A, Alqahtani H, Alshamrani M, Mahmoud E, Alothman A, Alsaedy A, Aldibasi O, Alhagan K, Asiri AM, AlJohani S, Al-Jeraisy M, Alaskar A. Multicentre randomised double-blinded placebo-controlled trial of favipiravir in adults with mild COVID-19. BMJ Open. 2021 Apr 14;11(4):e047495. doi: 10.1136/bmjopen-2020-047495. PMID 33853806